CLINICAL TRIAL: NCT07370870
Title: Is Cryotherapy Beneficial After Surgical Removal of Impacted Lower Third Molars? - A Randomized Split Mouth Clinical Trial
Brief Title: Is Cryotherapy Beneficial After Surgical Removal of Impacted Lower Third Molars?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henrique Tedesco (Other)
Responsible Party: Sponsor-Investigator, Henrique Tedesco, Sponsor-Investigator, Federal University of Rio Grande do Sul
Organization: Federal University of Rio Grande do Sul (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 75651517.4.0000.5347; 75651517.4.0000.5347 (Other: Universidade Federal do Rio Grande do Sul)
Record Dates: First submitted 2026-01-02; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cold Therapy
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: Randomized split-mouth clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (No Intervention): Patients in whom postoperative cryotherapy was not applied
- Group B (Experimental): Patients in whom postoperative cryotherapy was applied
  Interventions: Other: Cold Therapy

INTERVENTIONS:
Other: Cold Therapy — Postoperative cold therapy applied with ice packs
  Arms: Group B

SUMMARY:
The present study aimed to investigate the effects of cryotherapy on postoperative parameters (pain intensity, edema, trismus, and the quality of life) after lower third molar extraction. Patients underwent bilateral extraction of mandibular third molars in a single surgical procedure. Cryotherapy was applied to one side using facial ice packs, while no cryotherapy was performed on the contralateral side. Surgical procedures, postoperative instructions, and prescribed medications were identical for both sides. Consequently, the side treated with ice packs exhibited lower pain intensity, shorter pain duration, and reduced use of rescue medication.

ELIGIBILITY:
Inclusion Criteria

* Indication for bilateral surgical removal of mandibular third molars in similar positions
* Absence of systemic comorbidities
* Absence of local inflammatory processes
* Absence of local infectious processes
* No history of allergy to the prescribed medications
* No chronic use of antibiotics, anti-inflammatory drugs, corticosteroids, and/or analgesics

Exclusion Criteria

* Use of medications other than those prescribed by the surgeon
* Failure to provide the required data

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Effects of cryotherapy on postoperative pain intensity after lower third molar extraction - using a visual analog scale. | 7 days
  Evaluate the effects of cryotherapy on postoperative pain intensity following lower third molar extraction using a visual analog scale (VAS) ranging from 0 to 10, where 0 indicates no pain and 10 represents the worst pain imaginable. Pain intensity was recorded daily by the participants over a 7-day postoperative period.
Evaluate the effects of cryotherapy on postoperative edema after lower third molar extraction - using the mean of three linear facial measurements | 7 days
  Evaluate the effects of cryotherapy on postoperative edema following lower third molar extraction using three linear facial measurements: tragus to pogonion, tragus to oral commissure, and lateral canthus to the mandibular angle. Measurements were recorded in millimeters, and the mean of the three values was calculated to quantify edema. Assessments were performed preoperatively and postoperatively on the second and seventh days.
Evaluate the effects of cryotherapy on postoperative trismus after lower third molar extraction - measuring maximum mouth opening | 7 days
  Evaluate the effects of cryotherapy on postoperative trismus following lower third molar extraction by measuring maximum mouth opening. Patients were seated with the tragus-ala plane parallel to the ground. Measurements were obtained using a measuring tape and recorded in millimeters. Assessments were performed on postoperative days 0, 2, and 7.
Evaluate the effects of cryotherapy on postoperative quality of life after lower third molar extraction - using a questionnaire adapted from the Oral Health Impact Profile-14 (OHIP-14) | 7 days
  Evaluate the effects of cryotherapy on postoperative quality of life following lower third molar extraction using a questionnaire adapted from the Oral Health Impact Profile-14 (OHIP-14), consisting of 14 dichotomous (yes/no) questions addressing daily functional limitations. The questionnaire was administered on the day of surgery and completed by participants on postoperative days 0, 2, and 7.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-12-30): https://cdn.clinicaltrials.gov/large-docs/70/NCT07370870/Prot_SAP_ICF_000.pdf